CLINICAL TRIAL: NCT00845663
Title: Open Label, Randomized, Parallel Group, Single Dose, 2-way Comparison Bioequivalence Study of Certolizumab Pegol Solution Injected Either by a Pre-filled Syringe (Reference) or by an Auto-injection Device (Test) to Healthy Volunteers.
Brief Title: Comparison Bioequivalence Study: Pre-filled Syringe (Reference) Versus Auto-injection Device (Test)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C87045
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: certolizumab pegol; Cimzia; bioequivalence; Comparison Bioequivalence Study
MeSH Terms: interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-filled Syringe (Active Comparator): pre-filled syringe (reference)
  Interventions: Drug: Certolizumab pegol
- Auto-injection Device (Experimental): Auto-injection device (test)
  Interventions: Drug: Certolizumab pegol

INTERVENTIONS:
Drug: Certolizumab pegol — Auto-injection device (test) containing 1 mL of certolizumab pegol liquid formulation, 200 mg/mL; 2 injections
  Other Names: Cimzia®; CDP870; CZP
  Arms: Auto-injection Device
Drug: Certolizumab pegol — Pre-filled syringe (reference) containing 1 mL of certolizumab pegol liquid formulation, 200 mg/mL; 2 injections
  Other Names: Cimzia®; CDP870; CZP
  Arms: Pre-filled Syringe

SUMMARY:
To compare the bioavailability of a single 400 mg dose of certolizumab pegol solution (2 x 200mg subcutaneous injections) injected either by a pre-filled syringe (reference) or by an auto-injection device (test).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55 years.
* A Body mass Index (BMI) of 18 to 28 kg/m
* Good physical and mental health status determined on the basis of the medical history and a general clinical examination
* Electrocardiogram and clinical laboratory tests interpreted as "normal"
* QuantiFERON-TB test negative
* female subjects: medically accepted method of contraception

Exclusion Criteria:

* prohibited concomitant medication
* administered vaccines and immunoglobulins in the month preceding the certolizumab pegol injection
* history of significant disease, allergies
* history of drug and/or alcohol abuse
* hepatic enzyme inducing drug within 2 months before study drug administration
* any drugs having influence of the immune response and antibiotic in the month preceding the inclusion
* known to be intolerant to PEG
* previously received certolizumab pegol
* previously received an antibody product within 5-half lives of the antibody or within 3 months of the start of the study
* history of tuberculosis
* have serum hepatitis or is carrier of the Hepatitis B surface antigen (HBs Ag), or Hepatitis C antibody or who is HIV positive

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Rennes, France

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 159 subjects have been screened. Participant Flow presents all subjects randomized. Intent-to-treat and Safety population are identical to randomized population.
Groups:
- Pre-filled Syringe: Certolizumab pegol (CDP870) 400 mg pre-filled syringe (reference); syringe contains 1 mL of certolizumab pegol liquid formulation, 200 mg/mL ; 2 injections are given
- Auto-Injection Device: Certolizumab pegol (CDP870) 400 mg Auto injection device (test); Auto-injection device contains 1 mL of certolizumab pegol liquid formulation, 200 mg/mL ; 2 injections are given
Period: Overall Study
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Started | 49 | 49
Completed | 49 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-filled Syringe | Auto-Injection Device | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 49 | 98
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.78 (9.95) | 33.18 (9.63) | 35.98 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 24 | 21 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 48 | 49 | 97
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 49 | 49 | 98
Body Height [Mean (Standard Deviation); unit: cm] | 168.64 (9.47) | 170.12 (9.04) | 169.38 (9.24)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/square meter] | 23.36 (2.53) | 22.93 (2.43) | 23.15 (2.48)
Body Surface Area [Mean (Standard Deviation); unit: Square meter] | 1.759 (0.171) | 1.770 (0.172) | 1.765 (0.171)
Body Weight [Mean (Standard Deviation); unit: kilogram] | 66.59 (10.11) | 66.58 (10.23) | 66.59 (10.12)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Drug Concentration-time Curve From Time 0 to Infinity (AUC)
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Geometric Mean (Full Range); unit: microgram *day/mL
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
microgram *day/mL | 1308 [731 to 2364] | 1326 [691 to 2708]
Statistical Analysis 1: Comparison: Pre-filled Syringe vs Auto-Injection Device; Bioequivalence testing by using the 90% Confidence Interval; Test type: Non-Inferiority or Equivalence — Use of the 80-125 % bioequivalence range. If 90% confidence interval for ratio of geometric LS Means (percent) is included within these limits, the devices are considered bioequivalent; ANOVA; ANOVA for log-transformed values with treatment as factor has been used as the basis for calculation of estimated value and confidence interval; ratio of geometric LS Means (percent) = 101.33, 90% CI [92.84 to 110.58] — Ratio is Auto-injection device/Pre-filled syringe

2. Primary Outcome: Area Under the Plasma Drug Concentration-time Curve From Time 0 to the Last Quantifiable Point (AUC(0-t))
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Geometric Mean (Full Range); unit: microgram*day/mL
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
microgram*day/mL | 1269 [716 to 2293] | 1240 [592 to 2696]
Statistical Analysis 1: Comparison: Pre-filled Syringe vs Auto-Injection Device; Bioequivalence testing by using the 90% Confidence Interval; Test type: Non-Inferiority or Equivalence — Use of the 80-125% bioequivalence range. If 90% confidence interval for ratio of geometric LS Means (percent) is included within these limits, the devices are considered bioequivalent; ANOVA; ANOVA for log-transformed values with treatment as factor was taken as the basis for calculation of estimated value and confidence interval; ratio of geometric LS Means (percent) = 97.70, 90% CI [89.06 to 107.19] — Ratio is Auto-injection device/Pre-filled syringe

3. Primary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Geometric Mean (Full Range); unit: microgram/mL
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
microgram/mL | 61.6 [32.4 to 121.0] | 60.1 [29.1 to 105.0]
Statistical Analysis 1: Comparison: Pre-filled Syringe vs Auto-Injection Device; Bioequivalence testing by using the 90% Confidence Interval; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; ANOVA for log-transformed values with treatment as factor was taken as a basis for calculation of estimated value and the confidence interval; ratio of geometric LS Means (percent) = 97.54, 90% CI [87.33 to 108.94] — Ratio is Auto-injection device/Pre-filled syringe

4. Secondary Outcome: Time Point Where Log-linear Elimination Phase Begins (TLIN)
Description: TLIN describes timepoint for start of elimination phase determined on the basis of a linear regression model of the log-transformed concentration data.
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Median (Full Range); unit: days
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
days | 21.0 (9.05) [9.0 to 42.0] | 21.0 (8.89) [6.0 to 42.0]

5. Secondary Outcome: Lowest Quantifiable Concentration Time (LQCT)
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Median (Full Range); unit: days
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
days | 56.0 (16.3) [28.0 to 84.0] | 84.0 (17.0) [28.0 to 84.0]

6. Secondary Outcome: Apparent Terminal Elimination Rate Constant (λz)
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: 1/day
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
1/day | 0.0732 (0.0387) | 0.0639 (0.0189)

7. Secondary Outcome: Apparent Terminal Elimination Half-life (t1/2)
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Median (Full Range); unit: days
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
days | 10.9 [2.57 to 21.3] | 11.7 [5.99 to 24.1]

8. Secondary Outcome: Time Corresponding to Cmax (Tmax)
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Median (Full Range); unit: days
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
days | 5.00 [3.00 to 9.00] | 5.00 [2.04 to 14.0]

9. Secondary Outcome: Apparent Total Body Clearance (CL/F)
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Geometric Mean (Full Range); unit: mL/day
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
mL/day | 306 [169 to 547] | 302 [148 to 579]

10. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Geometric Mean (Full Range); unit: L
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
L | 4.58 [1.39 to 13.0] | 4.92 [2.07 to 10.9]

11. Secondary Outcome: Number of Subjects With Anti-certolizumab Pegol Antibody Plasma Level >2.4 Units/mL
Time Frame: After 12 and 24 hours, on day 3, 4, 5, 6, 7, 10, after week 2, 3, 4, 6, 8, 12
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants | 22 | 15

12. Secondary Outcome: Injection Pain Assessment on a Visual Analog Scale (VAS) Per Formulation and Per Time Point as Well as Change From Baseline (=Immediately After Injection) at One Hour After Injection
Description: Visual Analog Scale (VAS) ranges from 0 (no pain at all) to 100 mm (max. pain).
Time Frame: Immediately after injection and 1 hour after injection
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Units on a scale
  Immediately after injection | 28.9 (22.8) | 20.9 (15.6)
  1 hour after injection | 2.3 (4.0) | 1.1 (2.3)
  Change over time (1 hour after injection) | -26.6 (22.8) | -19.8 (15.6)

13. Secondary Outcome: Injection Questionnaire Per Formulation and Per Time Point - Afraid of Needles
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Before and 24 hours post-dose
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Before - not at all | 13 | 18
  Before - a little | 17 | 16
  Before - moderately | 17 | 14
  Before - very | 0 | 1
  Before - extremely | 1 | 0
  24 hours post-dose - not at all | 15 | 18
  24 hours post-dose - a little | 19 | 16
  24 hours post-dose - moderately | 14 | 14
  24 hours post-dose - very | 0 | 1
  24 hours post-dose - extremely | 1 | 0

14. Secondary Outcome: Injection Questionnaire Per Formulation and Per Time Point - Afraid of Having Injections
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Before and 24 hours post-dose
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Before - not at all | 11 | 13
  Before - a little | 21 | 17
  Before - moderately | 16 | 19
  Before - very | 0 | 0
  Before - extremely | 1 | 0
  24 hours post-dose - not at all | 13 | 13
  24 hours post-dose - a little | 21 | 17
  24 hours post-dose - moderately | 14 | 19
  24 hours post-dose - very | 0 | 0
  24 hours post-dose - extremely | 1 | 0

15. Secondary Outcome: Injection Site Reaction Questionnaire Per Formulation and Per Time Point - Pain
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Immediately after injection, 1 h and 24 h after injection
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Immediately after injection - not at all | 11 | 7
  Immediately after injection - a little | 16 | 26
  Immediately after injection - moderately | 18 | 13
  Immediately after injection - very | 4 | 2
  Immediately after injection - extremely | 0 | 1
  1 hour after injection - not at all | 35 | 32
  1 hour after injection - a little | 10 | 14
  1 hour after injection - moderately | 2 | 1
  1 hour after injection - very | 1 | 1
  1 hour after injection - extremely | 0 | 0
  24 hours after injection - not at all | 33 | 28
  24 hours after injection - a little | 9 | 16
  24 hours after injection - moderately | 5 | 1
  24 hours after injection - very | 1 | 2
  24 hours after injection - extremely | 1 | 0

16. Secondary Outcome: Injection Site Reaction Questionnaire Per Formulation and Per Time Point - Burning Sensation
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Immediately after injection, 1 hour and 24 hours after injection
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Immediately after injection - not at all | 23 | 23
  Immediately after injection - a little | 12 | 13
  Immediately after injection - moderately | 6 | 11
  Immediately after injection - very | 7 | 2
  Immediately after injection - extremely | 1 | 0
  1 hour after injection - not at all | 42 | 41
  1 hour after injection - a little | 4 | 8
  1 hour after injection - moderately | 1 | 0
  1 hour after injection - very | 1 | 0
  1 hour after injection - extremely | 1 | 0
  24 hours after injection - not at all | 39 | 38
  24 hours after injection - a little | 5 | 9
  24 hours after injection - moderately | 2 | 2
  24 hours after injection - very | 2 | 0
  24 hours after injection - extremely | 1 | 0

17. Secondary Outcome: Injection Site Reaction Questionnaire Per Formulation and Per Time Point - Cold Sensation
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Immediately after injection, 1 hour and 24 hours after injection
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Immediately after injection - not at all | 42 | 37
  Immediately after injection - a little | 6 | 11
  Immediately after injection - moderately | 1 | 1
  Immediately after injection - very | 0 | 0
  Immediately after injection - extremely | 0 | 0
  1 hour after injection - not at all | 47 | 49
  1 hour after injection - a little | 2 | 0
  1 hour after injection - moderately | 0 | 0
  1 hour after injection - very | 0 | 0
  1 hour after injection - extremely | 0 | 0
  24 hours after injection - not at all | 46 | 46
  24 hours after injection - a little | 3 | 3
  24 hours after injection - moderately | 0 | 0
  24 hours after injection - very | 0 | 0
  24 hours after injection - extremely | 0 | 0

18. Secondary Outcome: Injection Site Reaction Questionnaire Per Formulation and Per Time Point - Itching
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Immediately after injection, 1 hour and 24 hours after injection
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Immediately after injection - not at all | 46 | 44
  Immediately after injection - a little | 3 | 5
  Immediately after injection - moderately | 0 | 0
  Immediately after injection - very | 0 | 0
  Immediately after injection - extremely | 0 | 0
  1 hour after injection - not at all | 46 | 47
  1 hour after injection - a little | 3 | 2
  1 hour after injection - moderately | 0 | 0
  1 hour after injection - very | 0 | 0
  1 hour after injection - extremely | 0 | 0
  24 hours after injection - not at all | 47 | 46
  24 hours after injection - a little | 2 | 2
  24 hours after injection - moderately | 0 | 0
  24 hours after injection - very | 0 | 0
  24 hours after injection - extremely | 0 | 0

19. Secondary Outcome: Injection Site Reaction Questionnaire Per Formulation and Per Time Point - Redness
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Immediately after injection, 1 hour and 24 hours after injection
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Immediately after injection - not at all | 24 | 39
  Immediately after injection - a little | 19 | 8
  Immediately after injection - moderately | 6 | 2
  Immediately after injection - very | 0 | 0
  Immediately after injection - extremely | 0 | 0
  1 hour after injection - not at all | 28 | 47
  1 hour after injection - a little | 19 | 2
  1 hour after injection - moderately | 2 | 0
  1 hour after injection - very | 0 | 0
  1 hour after injection - extremely | 0 | 0
  24 hours after injection - not at all | 39 | 46
  24 hours after injection - a little | 10 | 3
  24 hours after injection - moderately | 0 | 0
  24 hours after injection - very | 0 | 0
  24 hours after injection - extremely | 0 | 0

20. Secondary Outcome: Injection Site Reaction Questionnaire Per Formulation and Per Time Point - Swelling
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Immediately after injection, 1 hour and 24 hours after injection
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Immediately after injection - not at all | 37 | 34
  Immediately after injection - a little | 11 | 14
  Immediately after injection - moderately | 1 | 1
  Immediately after injection - very | 0 | 0
  Immediately after injection - extremely | 0 | 0
  1 hour after injection - not at all | 39 | 40
  1 hour after injection - a little | 10 | 7
  1 hour after injection - moderately | 0 | 2
  1 hour after injection - very | 0 | 0
  1 hour after injection - extremely | 0 | 0
  24 hours after injection - not at all | 40 | 37
  24 hours after injection - a little | 8 | 11
  24 hours after injection - moderately | 1 | 1
  24 hours after injection - very | 0 | 0
  24 hours after injection - extremely | 0 | 0

21. Secondary Outcome: Injection Site Reaction Questionnaire Per Formulation and Per Time Point - Bruising
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Immediately after injection, 1 hour and 24 hours after injection
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Immediately after injection - not at all | 46 | 47
  Immediately after injection - a little | 3 | 2
  Immediately after injection - moderately | 0 | 0
  Immediately after injection - very | 0 | 0
  Immediately after injection - extremely | 0 | 0
  1 hour after injection - not at all | 49 | 47
  1 hour after injection - a little | 0 | 2
  1 hour after injection - moderately | 0 | 0
  1 hour after injection - very | 0 | 0
  1 hour after injection - extremely | 0 | 0
  24 hours after injection - not at all | 45 | 46
  24 hours after injection - a little | 4 | 3
  24 hours after injection - moderately | 0 | 0
  24 hours after injection - very | 0 | 0
  24 hours after injection - extremely | 0 | 0

22. Secondary Outcome: Injection Site Reaction Questionnaire Per Formulation and Per Time Point - Hardening
Description: Categorized answer ranges from not at all to extremely.
Time Frame: Immediately after injection, 1 hour and 24 hours after injection
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Number analyzed (Participants) | 49 | 49
Participants
  Immediately after injection - not at all | 37 | 34
  Immediately after injection - a little | 11 | 12
  Immediately after injection - moderately | 1 | 2
  Immediately after injection - very | 0 | 1
  Immediately after injection - extremely | 0 | 0
  1 hour after injection - not at all | 38 | 34
  1 hour after injection - a little | 9 | 12
  1 hour after injection - moderately | 2 | 3
  1 hour after injection - very | 0 | 0
  1 hour after injection - extremely | 0 | 0
  24 hours after injection - not at all | 38 | 38
  24 hours after injection - a little | 11 | 10
  24 hours after injection - moderately | 0 | 1
  24 hours after injection - very | 0 | 0
  24 hours after injection - extremely | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pre-filled Syringe | Auto-Injection Device
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/49
Other Adverse Events (participants affected / at risk) | 30/49 | 31/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-filled Syringe (N=49) | Auto-Injection Device (N=49)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-filled Syringe (N=49) | Auto-Injection Device (N=49)
Abdominal Pain (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 6
Asthenia (General disorders) | 3 | 1
Influenza like illness (General disorders) | 0 | 5
Nasopharyngitis (Infections and infestations) | 10 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 22 | 19
Dysmenorrhoea (Reproductive system and breast disorders) | 4 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.